CLINICAL TRIAL: NCT06354179
Title: Evaluation of the Benefits of Administering Immunosuppressive Drugs as Single Daily Doses Over the First Year After Liver Transplantation
Brief Title: Evaluation of the Benefits of Administering Immunosuppressive Drugs as Single Daily Doses Over the First Year After Liver Transplantation (EASY)
Acronym: EASY
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 87RI23_0031 (EASY)
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Liver Transplantation; Immunosuppression
Keywords: liver transplantation; immunosuppression; tacrolimus; mycophenolate; adherence; once-daily intake

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard of care 1 (Active Comparator)
  Interventions: Drug: XR-tacrolimus QD + MMF BID
- Test 1 (Experimental)
  Interventions: Drug: XR-tacrolimus QD + MMF BID then MMF QD
- Test 2 (Experimental)
  Interventions: Drug: LCP-tacrolimus QD + MMF QD then MMF QD
- Standard of care 2 (Active Comparator)
  Interventions: Drug: LCP-tacrolimus QD + MMF BID

INTERVENTIONS:
Drug: XR-tacrolimus QD + MMF BID then MMF QD — Patients start on XR-Tacrolimus once daily (QD) and MMF twice daily (BID) as per the usual care. At 6 months post-transplantation (±1 month) MMF administration frequency will be switched from BID to QD, in the morning, at the same daily dose
  Arms: Test 1
Drug: XR-tacrolimus QD + MMF BID — Patients receive XR-tacrolimus once daily (QD) and MMF twice daily (BID) as per the usual care.
  Arms: Standard of care 1
Drug: LCP-tacrolimus QD + MMF QD then MMF QD — Patients start on LCP-Tacrolimus once daily (QD) and MMF twice daily (BID) as per usual care. At 6 months post-transplantation (±1 month), MMF administration frequency will be switched from BID to QD, in the morning, at the same daily dose
  Arms: Test 2
Drug: LCP-tacrolimus QD + MMF BID — Patients receive LCP-tacrolimus once daily (QD) and MMF twice daily (BID) as per the usual care.
  Arms: Standard of care 2

SUMMARY:
World Health Organization considers non-adherence has a strong negative impact on the health of patients with chronic diseases. In transplantation, adherence to immunosuppressive drug regimens associates with late rejection and graft loss making it a critical determinant of patient outcome. The prevalence of non-adherence in transplant patients, including liver transplant patients, can be as high as 40%. Among others, life-long intake and complexity of immunosuppressive regimen make patients prone to non-adherence. For instance, non-adherence is more prevalent among patients with higher numbers of immunosuppressive drugs. One of the most commonly cited causes of non-adherence is forgetfulness and disruptions in routine, with the evening dose of twice daily regimens being the most likely to be affected6. Besides non-adherence, the constraints generated in everyday life by immunosuppression (including timely and regular drug intake) and the complexity of the immunosuppressive regimens represent a burden for the patients and are probably associated with a health-related quality of life deterioration. Therefore, long-term adherence and quality of life after liver transplantation might be improved by using a well-tolerated and easy-to-handle immunosuppressive regimen.

The immunosuppressive regimen after liver transplantation is in most cases based on different combinations of tacrolimus, mycophenolate mofetil and corticosteroids. While corticosteroids are administered once daily, tacrolimus can be administered either twice-daily (BID) as an immediate-release, or once-daily (QD) as an extended-release formulation. Among once-daily tacrolimus formulations, LCP-tacrolimus (ENVARSUS XR®) is approved for the prevention of transplant rejection in adult liver allograft recipients. It has demonstrated similar outcomes compared to immediate-release tacrolimus BID, in both kidney and liver transplantation. Mycophenolate has only been approved for BID administration, preventing from taking all immunosuppressive drugs once daily. Yet, single daily dosing would probably contribute to better adherence and quality of life in patients receiving a life-long treatment.

Although the half-life of mycophenolic acid (MPA), the active moiety of mycophenolate mofetil (MMF) is compatible with once-daily administration, no published randomized clinical study has ever evaluated the efficacy and safety of MMF administered QD.

The narrow therapeutic index and wide pharmacokinetic variability of tacrolimus and mycophenolate justify individual dose adjustment by means of therapeutic drug monitoring (TDM), in order to minimize the risk of acute rejection and the occurrence of adverse events. For tacrolimus, TDM is generally based on the trough concentration (C0) and sometimes on the area under the concentration-time curve (AUC), while for mycophenolate it should be based on the AUC of MPA. However, the dose adjustment of MMF in liver transplant patients is most of the time performed a posteriori, based on clinical signs of inefficacy of toxicity.

Limited sampling strategies with maximum a posteriori Bayesian estimation have been developed by our team for both molecules in adult liver transplant patients to estimate their AUC, which is considered the best marker of exposure for both. Therefore, tacrolimus AUC0-24h can be estimated by Bayesian estimation using samples collected before administration (C0), 8 (C8h) and 12 (C12h) hours after the administration of ENVARSUS XR®, or 1 and 3 hours after the administration of PROGRAF® and ADVAGRAF®. For mycophenolate, the MPA AUC can be estimated using samples collected 20 min, 1 and 3 hours after MMF administration, by Bayesian estimation.

Even if limited to 2 or 3 blood samples, tacrolimus TDM for ENVARSUS® requires late sampling (12h post-dose). To overcome the necessity of a longer hospital stay, microsampling devices (MSD) such as the Volumetric absorptive microsampling (VAMS®) device (Mitra®) can be used by the patients to take samples themselves, at home. Moreover, they are less invasive than venipuncture and collect low but accurate volumes of blood for analysis.

In this context, we propose a randomized controlled non-inferiority study to demonstrate that in liver transplant recipients, an immunosuppressive strategy based on single daily doses of LCP-tacrolimus (ENVARSUS XR®) and mycophenolate mofetil (CELLCEPT®) started at M6 post-transplantation is not inferior to XR-tacrolimus (ADVAGRAF®) and MMF administered BID, in terms of incidence of treatment failure (see below) at the end of the first year after transplantation, and to obtain adherence, quality of life and safety data. In order to compare solely MMF QD to MMF BID, patients on ENVARSUS XR® and MMF QD will be compared to a third group of patients receiving ENVARSUS XR® and MMF BID. A direct comparison of efficacy and safety, quality of life, adherence and exposure indices will be performed between ENVARSUS XR® and ADVAGRAF®.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of a first liver allograft from a deceased donor
* Transplanted for less than four weeks at enrolment.
* Without inter-current progressive life-threatening or graft-threatening disease.
* Having signed a written informed consent for their participation in the study.
* Affiliated to, or beneficiary of, a social security regimen

Exclusion Criteria:

* Recipients of a split-liver transplantation.
* Recipients of any transplanted organ other than the liver
* Patient who has undergone colon resection
* Patients under legal protection (guardianship, curatorship).
* Patient presenting any contra-indication to tacrolimus or to MMF according to the summary of product characteristics (SmPC) of ENVARSUS®, ADVAGRAF® and CELLCEPT®.
* Patients in whom everolimus-based calcineurin inhibitors (CNI) minimization is anticipated
* Patients treated with HIV or HCV protease inhibitors.
* Pregnant or lactating women.
* Women of childbearing potential without any effective contraceptive method (according to the guidelines of CTFG, Clinical Trial Facilitation Group, related to contraception and pregnancy test in clinical trials) or not practicing sexual abstinence.
* Sexually active men having a female partner, without any effective contraception.
* Patients incapable of understanding the purposes and risks of the study, who cannot give written informed consent, or who are unwilling to comply with the study protocol.
* Patients enrolled in another clinical study evaluating drugs or therapeutic strategies potentially interfering with the objectives of the EASY study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2028-04-15 (Estimated); Study Completion 2028-04-15 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | month 12
  Treatment failure, defined by the occurrence of any of the following events: Patient death, Graft loss, Biopsy-proven acute rejection, rejection activity index score ≥4 according to the Banff criteria

SECONDARY OUTCOMES:
Adherence to treatment | Month 18
  Adherence evaluated using the BAASIS questionnaire and patient diaries. Arm LCP-tacrolimus vs. Arm XR-tacrolimus
measuring of quality of life | Month 18
  Health-related quality of life composite scores evaluated using the SF-36 questionnaire. Arm LCP-tacrolimus vs. Arm XR-tacrolimus
Adherence to treatment | Month 18
  Adherence evaluated using the BAASIS questionnaire and patient diaries. Benefits of switching from Arm MMF BID to Arm MMF QD
measuring of quality of life | Month 18
  Health-related quality of life composite scores evaluated using the SF-36 questionnaire. Benefits of switching from Arm MMF BID to Arm MMF QD
Appearance Adverse events | month 18
  Adverse events and their severity whenever applicable during the first year after transplantation ( Gastro-intestinal, Cytomegalovirus (CMV) infection or reactivation, Neutropenia, Sepsis, Renal function impairment, post-transplant diabetes mellitus, Hypertension, Hyperlipidemia, Tremor). Arm LCP-tacrolimus vs. Arm XR-tacrolimus
Appearance Adverse events | month 18
  Adverse events and their severity whenever applicable during the first year after transplantation ( Gastro-intestinal, CMV infection or reactivation, Neutropenia, Sepsis, Renal function impairment, post-transplant diabetes mellitus, Hypertension, Hyperlipidemia, Tremor). Arm MMF BID to Arm MMF QD
Comparison tacrolimus daily exposure | month 18
  average daily exposure of tacrolimus by AUC 0-24h determined by Bayesian estimation compare between the 3 arms
Comparison of MPA daily exposure | month 18
  average daily exposure of MPA AUC 0-24h determined by Bayesian estimation compare between the 3 arms
Comparison of Tacrolimus dose | month 18
  measurement of Tacrolimus dose at C0 to comparison between the 3 arms
Comparison of Tacrolimus AUC 0-24h | month 18
  measurement of Tacrolimus AUC 0-24h to comparison between the 3 arms
Comparison of MPA AUC 0-24h | month 18
  measurement of MPA AUC 0-24h to comparison between the 3 arms

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - CHU de Besançon - Hôpital Jean Minjoz, Besançon
  - Beaujon hospital - APHP, Clichy
  - CHU de Dijon Bourgogne, Dijon
  - Lille university hospital, Lille
  - Limoges university hospital, Limoges
  - Lyon university hospital, Lyon
  - APHP, Marseille
  - Montpellier university hospital, Montpellier
  - Nice university hospital, Nice
  - Pitie Salpetriere hospital - APHP, Paris
  - Bordeaux university hospital, Pessac
  - Poitiers university hospital, Poitiers
  - Rennes university hospital, Rennes
  - Strasbourg university hospital, Strasbourg
  - Toulouse university hospital, Toulouse
  - Tours university Hospital, Tours
  - Paul Brousse Hospital - APHP, Villejuif

IPD SHARING:
Plan to Share IPD: No